CLINICAL TRIAL: NCT05729529
Title: Impact of Alpha Lipoic Acid Efficacy in Burning Mouth Syndrome Using a Topical Gel
Brief Title: Impact of Alpha Lipoic Acid Efficacy in Burning Mouth Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-20
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome

STUDY DESIGN:
Intervention Model Description: The main objective of this study was to evaluate the efficacy of lipoic acid over placebo in the management of BMS
Who Masked: Participant, Investigator
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipoic acid gel (Active Comparator): Patients were treated with a topic gel of lipoic acid
  Interventions: Other: Lipoid acid gel
- Placebo (Placebo Comparator): Patients treated with a placebo gel control
  Interventions: Drug: Placebo

INTERVENTIONS:
Other: Lipoid acid gel — Topic lipoid acid gel used with topic oral gel used on tongue
  Arms: Lipoic acid gel
Drug: Placebo — Placebo oral gel used on tongue
  Arms: Placebo

SUMMARY:
A double-blind placebo-controlled trial is conducted in order to evaluate the efficacy of alpha lipoic acid (ALA) and determine the statistical significance of the outcome variables. Burning mouth syndrome (BMS) is defined as an oral burning sensation in the absence of clinical signs which could justify the syndrome.

Recent studies suggest the existence of neurological factors as a possible cause of the disease.

DETAILED DESCRIPTION:
A double-blind placebo-controlled trial is conducted in order to evaluate the efficacy of alpha lipoic acid (ALA) and determine the statistical significance of the outcome variables.

60 patients with BMS, in two groups: case group with 600 mg/day and placebo as control group; with a follow-up of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with BMS who reported a history of continuous oral burning pain for more than 4 months with no clinical signs that could justify the syndrome

Exclusion Criteria:

* clinically diagnosed with BMS who reported a history of continuous oral burning pain for more than 4 months with no clinical signs that could justify the syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-05-25 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of burning mouth | 6 months
  Evolution of burning mouth symptoms change through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Time Frame: 1 year
Access Criteria: Pubmed